CLINICAL TRIAL: NCT02989168
Title: A Phase II Open Label Study to Evaluate the Effect of GBT440 on Hypoxemia in Subjects With Idiopathic Pulmonary Fibrosis (IPF) Who Are Using Supplemental Oxygen at Rest (ZEPHYR)
Brief Title: Study to Evaluate the Effect of GBT440 Administered to Subjects With IPF on Supplemental Oxygen at Rest
Acronym: Zephyr
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated due to lack of clinically meaningful benefit
Sponsor: Global Blood Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: GBT440-026
Record Dates: First submitted 2016-11-28; First posted 2016-12-12 (Estimated); Results first posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-07

CONDITIONS: Idiopathic Pulmonary Fibrosis; Hypoxemia
Keywords: Idiopathic pulmonary fibrosis; hypoxemia; oxygen
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Hypoxia | interventions — voxelotor

ARMS (2):
- GBT440 900 mg Dose (Experimental): Part A, 900 mg
  GBT440: Capsules which contain GBT440 drug substance in Swedish orange
  Interventions: Drug: GBT440
- GBT440 1500 mg Dose (Experimental): Part B , 1500 mg
  GBT440: Capsules which contain GBT440 drug substance in Swedish orange
  Interventions: Drug: GBT440

INTERVENTIONS:
Drug: GBT440 — GBT440: Capsules which contain GBT440 drug substance in Swedish orange

SUMMARY:
This is an open label study in which eligible IPF subjects who are using supplemental oxygen at rest will receive GBT440 orally daily.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of IPF.
* Receiving supplemental oxygen for use at rest.
* Weight ≥ 40 kg.
* Male or female of child bearing potential willing and able to use highly effective methods of contraception from study start to 30 days after the last dose of study drug.

Exclusion Criteria:

* FEV1/FVC < 70%
* History of other interstitial lung diseases.
* Subject plans to begin or has commenced pulmonary rehabilitation within 30 days of screening.
* Corticosteroid (> 10 mg per day of prednisone or an equivalent) administered for 7 days or longer, within 30 days of screening.
* Participated in another clinical trial of an investigational drug (or medical device) within 30 days or 5-half-lives, whichever is longer, prior to screening, or is currently participating in another trial of an investigational drug (or medical device).
* Female who is breast-feeding or pregnant
* Current smoker or history of smoking within 3 months from screening

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-11; Primary Completion 2017-10-23 (Actual); Study Completion 2017-10-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (6):
  - Birmingham, Alabama
  - Denver, Colorado
  - New Orleans, Louisiana
  - Philadelphia, Pennsylvania
  - Nashville, Tennessee
  - Salt Lake City, Utah
- United Kingdom (3):
  - London
  - Manchester
  - Southampton

RESULTS

PARTICIPANT FLOW:
Groups:
- GBT440 900 mg Dose: Part A , 900 mg daily dose
  GBT440: Capsules which contain GBT440 drug substance in Swedish orange
- GBT440 1500 mg Dose: Part B , 1500 mg daily dose
  GBT440: Capsules which contain GBT440 drug substance in Swedish orange
Period: Overall Study
Arm/Group | GBT440 900 mg Dose | GBT440 1500 mg Dose
Started | 11 | 3
Completed | 7 | 0
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Adverse Event | 1 | 2
Not completed — Sponsor stopped study. | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- GBT440 900 mg Dose: Part A, 900 mg daily dose
  GBT440: Capsules which contain GBT440 drug substance in Swedish orange
- GBT440 1500 mg Dose: Part B, 1500 mg daily dose
  GBT440: Capsules which contain GBT440 drug substance in Swedish orange
- Total: Total of all reporting groups
Arm/Group | GBT440 900 mg Dose | GBT440 1500 mg Dose | Total
Number analyzed (Participants) | 11 | 3 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (6.12) | 70.3 (5.69) | 68.7 (5.88)
Age, Continuous [Median (Full Range); unit: years] | 69.0 [59 to 77] | 72.0 [64 to 75] | 70.0 [59 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 10 | 2 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 3 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 3 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Oxygen Saturation at End of Treatment Period Compared to Baseline
Time Frame: Days 1 to 90
Population: Since study was stopped prematurely, complete data for all participants were not analyzable so no efficacy results are presented.
Groups:
- GBT440 900 mg Dose: Part A
  GBT440: Capsules which contain GBT440 drug substance in Swedish orange
- GBT440 1500 mg Dose: Part B
  GBT440: Capsules which contain GBT440 drug substance in Swedish orange
Arm/Group | GBT440 900 mg Dose | GBT440 1500 mg Dose
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Supplemental Oxygen Requirement at End of Treatment Period Compared to Baseline
Time Frame: Days 1 to 90
Population: as for outcome 1
Arm/Group | GBT440 900 mg Dose | GBT440 1500 mg Dose
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Evaluate the Effect of GBT440 on Resting and Post-exercise Alveolar-arterial O2 Tension Difference [P(A-a) O2] at End of Treatment Period Compared to Baseline
Time Frame: Days 1 to 90
Population: as for outcome 1
Arm/Group | GBT440 900 mg Dose | GBT440 1500 mg Dose
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Evaluate the Effect of GBT440 on Performance of the 6MWT
Time Frame: Days 1 to 90
Population: as for outcome 1
Arm/Group | GBT440 900 mg Dose | GBT440 1500 mg Dose
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Evaluate the Effect of GBT440 on IPF Related Symptoms Using Patient Related Outcomes
Time Frame: Days 1 to 90
Population: as for outcome 1
Arm/Group | GBT440 900 mg Dose | GBT440 1500 mg Dose
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Evaluate Pulmonary Function Using Pulmonary Function Tests (FVC and DLco)
Description: Spirometry measurements will include forced vital capacity (FVC) and diffusing capacity of the lung for carbon monoxide (DLco).
Time Frame: Days 1 to 90
Population: as for outcome 1
Arm/Group | GBT440 900 mg Dose | GBT440 1500 mg Dose
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.0
Time Frame: Days 1 to 90
Population: Participant had at least one dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | GBT440 900 mg Dose | GBT440 1500 mg Dose
Number analyzed (Participants) | 11 | 3
Participants | 11 | 3

8. Secondary Outcome: Pharmacokinetic Parameters of GBT440 in Plasma and Whole Blood (Minimum Concentration (Cmin))
Description: PK parameters of GBT440 administered daily orally for 90 days in plasma and whole blood, including but not limited to, minimum concentration (Cmin), at steady state.
Time Frame: Day 1 (15 mins post-dose and 2-4h post-dose), Day 15 (pre-dose), Day 30 (pre-dose), Day 60 (pre-dose and 2-4h post-dose), Day 90 (pre-dose), Day 105 (during study visit), and Day 120 (during study visit)
Population: Complete PK data were not analyzable for any participant.
Arm/Group | GBT440 900 mg Dose | GBT440 1500 mg Dose
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Screening to 90 days
Arm/Group | GBT440 900 mg Dose | GBT440 1500 mg Dose
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/3
Serious Adverse Events (participants affected / at risk) | 3/11 | 2/3
Other Adverse Events (participants affected / at risk) | 11/11 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GBT440 900 mg Dose (N=11) | GBT440 1500 mg Dose (N=3)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GBT440 900 mg Dose (N=11) | GBT440 1500 mg Dose (N=3)
Atrial flutter (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Fatigue (General disorders) | 3 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 1 | 0
Hepatic mass (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Viral sinusitis (Infections and infestations) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Since this study was stopped prematurely, no efficacy results will be presented.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2017-06-05): https://cdn.clinicaltrials.gov/large-docs/68/NCT02989168/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/68/NCT02989168/SAP_001.pdf